CLINICAL TRIAL: NCT00777504
Title: Study to the Optimal Duration of Therapy With Oral Angiogenesis Inhibitors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO200801
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Renal Cell Carcinoma; Gastrointestinal Stromal Tumor
Keywords: angiogenesis; inhibitor; duration of therapy; GIST
MeSH Terms: conditions — Carcinoma, Renal Cell; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): When PD is being determined the patient will continue with the oral angiogenesis inhibitors for 2 more weeks. After 2 weeks, an Avastinscan will be made and/or a dynamic contrast enhanced MRI (DCE-MRI). After evaluating these scans patients in group A now stop the orale angiogenesis inhibitor.
  Interventions: Drug: usage oral angiogenesis inhibitor
- B (Active Comparator): When PD is being determined the patient will continue with the oral angiogenesis inhibitors for 2 more weeks. After 2 weeks, an Avastinscan will be made and/or a dynamic contrast enhanced MRI (DCE-MRI). After evaluating these scans patients in group B continue with angiogenesis inhibitors for 2 more weeks. After these 2 weeks(so 4 weeks after inclusion) another Avastinscan will be made and/or a dynamic contrast enhanced MRI (DCE-MRI) and a FDG-PET-scan.
  Interventions: Drug: stop oral angiogenesis inhibitor

INTERVENTIONS:
Drug: usage oral angiogenesis inhibitor — see under 'study arms'
  Arms: A
Drug: stop oral angiogenesis inhibitor — see under 'study arms'
  Arms: B

SUMMARY:
The purpose of this study is to determine if and how often an unexpected fast increase of disease and complaints shows after stopping the anti-angiogenetic therapy

DETAILED DESCRIPTION:
Until now, in trials it is common to stop therapy when progressive disease occurs; RECIST criteria are used, in which progressive disease is defined as >20% increase of the sum of the longest diameter of the lesions, or occurence of new lesions. However, angiogenesis inhibitors have a rather cytostatic than cytotoxic effect compared to chemotherapeutics, as a result of which less frequently reduction of tumor volume is being seen.

Often in the centre of the lesion necrosis is shown. Sometimes accompanied with edema; so even tumor volume increase can be the result without real progression being the case. Recently, in our clinic, we found a number of patients, treated with oral angiogenesis inhibitors, a remarkable quickening of progressive disease and complaints after stopping this treatment. Reintroduction of the same or another type of angiogenesis inhibitor subsequently lead to a new stabilization. The causality of this phenomenon is unknown. Perhaps that the inhibitory effect of the angiogenesis is not fully exhausted at the moment that progressive disease on CT is observed. An alternative explanation is contra reaction of longterm angiogenetic inhibition through upregulation of proangiogenic factors with subsequent vascular expansion and edema. This study means to gain more insight information about the optimal treatment policy when progressive disease is found in patients treated with oral angiogenesis inhibitors. Because of the increase of patients that is being treated with these products, both in trials as in daily clinical practice, this is important to investigate.

ELIGIBILITY:
Inclusion Criteria:

* metastatic or advanced solid cancer that is treated with an oral angiogenesis inhibitor, with clinical indication to stop this therapy based on progressive disease as defined by the RECIST criteria on the CT scan. It needs a minimum of 1 previous evaluation of stable disease and the patient must have been treated with angiogenesis inhibitors for at least 12 weeks.
* age ≥18 years
* given informed consent

Exclusion Criteria:

* pregnant or lactating
* metastatic sites solely in bone or liver
* contraindication for CT or Avastin scan (claustrophobia, severe renal function disorder, allergy for contrast fluids, allergy for Avastin)
* insufficient condition to continue treatment with angiogenesis inhibitors.
* contraindication for dynamic contrast MRI (deteriorated renal functions with clearance <60ml/min, metal in body, claustrophobia, pacemaker, defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-01 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Signs of progressive disease on CT-scan, DCE-MRI or Avastin scan | 4 weeks

SECONDARY OUTCOMES:
Effect on Quality of life as record by questionaires | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Medical Center Nijmegen st Radboud, Nijmegen, Gelderland, Netherlands